CLINICAL TRIAL: NCT03691844
Title: A Placebo-controlled, Double-blind, Randomized, Trial of AMZ001 for the Treatment of Knee Osteoarthritis Symptoms
Brief Title: AMZ001 for the Treatment of Knee Osteoarthritis Symptoms
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Amzell (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMZ001-006
Record Dates: First submitted 2018-09-18; First posted 2018-10-02 (Actual); Results first posted 2020-10-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Osteoarthritis, Knee
Keywords: AMZ001
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: placebo-controlled, double-blind, randomized, parallel study
Who Masked: Participant, Investigator
Masking Description: 3 treatment arms will be double-blind, the 4th (comparator) will be single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AMZ001 + Placebo (Experimental): on the target knee
  Interventions: Drug: AMZ001
- AMZ001 (Experimental): on the target knee
  Interventions: Drug: AMZ001
- Placebo (Placebo Comparator): on the target knee
  Interventions: Drug: Placebo
- Comparator (Active Comparator): Diclofenac gel on the target knee
  Interventions: Drug: Comparator

INTERVENTIONS:
Drug: AMZ001 — diclofenac gel
  Arms: AMZ001; AMZ001 + Placebo
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Comparator — diclofenac gel
  Other Names: active comparator
  Arms: Comparator

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel group, 4-week trial of a formulation of AMZ001 once or twice daily versus placebo twice daily, including a single-blind treatment group with a commercial gel four times daily.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel group, 4-week trial of a formulation of AMZ001 once or twice daily versus placebo twice daily, including a single-blind treatment group with a commercial gel four times daily. Participants will be evaluated for osteoarthritis by X-ray images of the knees and one knee will be selected for treatment as the target knee. The study gel will be applied directly to that knee throughout the 4 weeks of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Osteoarthritis of the knee, according the American College of Rheumatology (ACR) clinical and X-ray criteria.
2. Pain score rated on an 11-point numerical rating scale of the target knee of ≥ 20 and ≤ 45 out of 50 in response to the WOMAC pain sub-score (5 questions), at the time of screening, after washout of any pain relief medication.
3. Women of child-bearing potential must use at least an acceptably effective method of contraception from enrollment up to at least 3 months after the study end.
4. Knee pain in the target knee for 14 days of the preceding month (knee pain due to osteoarthritis and not due to another condition such as bursitis, tendinitis, etc.) based on subject report.
5. On stable pain therapy (i.e., at least 3 days per week for the previous month) with an oral or topical NSAID prescribed by physician for 30 days prior to the Screening Visit and/or prescribed over-the-counter.
6. Except for osteoarthritis, in reasonably good health as determined by the Investigator.

Exclusion Criteria:

1. Known or suspected hypersensitivity to diclofenac, other non-steroidal anti-inflammatory drugs or related substances including aspirin, any of the components in either of the investigation products, or any physical impediment to gel application on the target knee.
2. Injection of corticosteroids or hyaluronic acid in the target knee within 6 months of screening or into any other joint within 30 days of screening.
3. High dose oral/injected corticosteroid treatment of more than 14 days during the past 6 months prior to screening.
4. Major surgery or arthroscopy of the target knee within the previous year prior to screening.
5. Planned surgery of the target knee within the next 3 months.
6. Presence of an additional non-osteoarthritic disease affecting either knee, such as rheumatoid arthritis, psoriasis, gout or pseudo-gout, if there is reason to believe that the disease(s) may significantly interfere with the interpretation of the clinical response to the study drug.
7. Medical history of coronary artery bypass graft surgery.
8. Current cancer or treatment for cancer within the past five years, with the exception of non-melanoma skin cancer, unless affecting the target knee area.
9. Secondary osteoarthritis of the target knee, previous procedures or trauma affecting joint of the target knee.
10. Reported incidence of any of the following diseases: known osteoarthritis of the hip(s) if pain in hip(s) exceeds that of the target knee using the WOMAC Hip Pain subscore, presence of significant back pain, or at least one migraine attack within the past 12 months before screening, as reported by the subject.
11. Body Mass Index > 45.0 kg/m2.
12. Generalized skin irritation, previous skin reactions upon use of topical NSAIDs, current skin irritation or redness at the planned site of gel application, or significant skin disease including psoriasis, as judged by the investigator.
13. Known presence of a ulcer or any gastrointestinal bleeding within 6 months prior to screening.
14. Use of moderate or higher doses of opioid medication for the treatment of pain within 6 weeks before the screening visit.
15. Use of duloxetine, pregabalin, or gabapentin within 4 weeks before the screening visit.
16. History of alcohol or drug abuse within the past year prior to randomization.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (3):
  - Clinical Research Consulting, Milford, Connecticut
  - Premier Medical Associates, The Villages, Florida
  - Upstate Clinical Research Associates, Williamsville, New York
- Czechia (3):
  - CCR Brno, s.r.o, Brno
  - CCR Czech, a.s, Pardubice
  - CCR Prague s.r.o., Prague
- Sanos Clinic, Herlev, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seven trial sites in Denmark (1 site), Czech Republic (3 sites) and the USA (3 sites).
  Trial initiation: 04-Oct-2018 Trial completion: 09-Jul-2019
Groups:
- AMZ001 BID: on the target knee
  AMZ001 gel twice daily.
  BID: Twice a day
- AMZ001 + Placebo QD: on the target knee
  AMZ001 gel once daily, Placebo gel once daily.
  QD: Every day/daily
- Placebo BID: on the target knee
  Placebo gel twice daily.
  BID: twice a day/ twice daily
- Voltaren 1% QID: on the target knee
  Voltaren gel 1% applied 4 times a day
  QID: 4 times every day
Period: Overall Study
Arm/Group | AMZ001 BID | AMZ001 + Placebo QD | Placebo BID | Voltaren 1% QID
Started | 121 | 121 | 121 | 81
Completed | 114 | 109 | 108 | 70
Not Completed | 7 | 12 | 13 | 11

BASELINE CHARACTERISTICS:
Groups:
- AMZ001 BID: on the target knee
  AMZ001 gel twice daily.
  BID: twice a day/twice daily
- Placebo BID: on the target knee
  Placebo gel twice daily.
  BID: 2 times a day/ twice a day
- Voltaren 1% QID: on the target knee
  Voltaren gel 1% applied 4 times a day
- Total: Total of all reporting groups
Arm/Group | AMZ001 BID | AMZ001 + Placebo QD | Placebo BID | Voltaren 1% QID | Total
Number analyzed (Participants) | 121 | 121 | 121 | 81 | 444
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 60 | 55 | 62 | 39 | 216
  >=65 years | 61 | 66 | 59 | 42 | 228
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 83 | 77 | 54 | 297
  Male | 38 | 38 | 44 | 27 | 147
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 3 | 1 | 5
  Not Hispanic or Latino | 120 | 121 | 118 | 80 | 439
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 6 | 1 | 4 | 3 | 14
  White | 115 | 119 | 115 | 77 | 426
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Baseline WOMAC pain sub-score [Mean (Standard Deviation); unit: score on a scale] — Baseline scores in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain sub-score (questions 1-5; score 0 [no pain]-50 [extreme pain]) on target knee. The WOMAC scores were normalized to a 0-100 point scale for data analysis, where higher scores indicates greater pain.
  score on a scale | 28.2 (6.07) | 27.5 (5.24) | 27.1 (4.82) | 27.3 (5.48) | 27.5 (5.41)

OUTCOME MEASURES:

1. Primary Outcome: WOMAC Pain Sub-score
Description: Change from baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain sub-score (questions 1-5; score 0 [no pain]-50 [extreme pain]) on target knee. The WOMAC scores were normalized to a 0-100 point scale for data analysis, where higher scores indicate greater pain, stiffness or difficulty in performing daily tasks.
Time Frame: baseline, week 4
Population: The mITT (modified Intent to treat; N=120) population set includes subjects with a baseline and at least one post-treatment WOMAC pain sub-score and was used in statistical analysis for primary and secondary endpoint outcome measures.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- AMZ001 BID: AMZ001 gel twice daily
- AMZ001 + Placebo QD: on the target knee
  AMZ001 gel once daily, Placebo gel once daily.
- Placebo BID: Placebo gel twice daily
Arm/Group | AMZ001 BID | AMZ001 + Placebo QD | Placebo BID
Number analyzed (Participants) | 120 | 120 | 120
score on a scale | -26.49 [-29.6 to -23.38] | -27.33 [-30.5 to -24.17] | -22.73 [-25.90 to -19.55]

2. Secondary Outcome: WOMAC Total Score and WOMAC Function and Stiffness
Description: Change from baseline in Western Ontario McMasters Universities Osteoarthritis Index (WOMAC) total score and WOMAC function (degree of difficulty experienced in performing daily activities - 17 questions score 0-170) and stiffness (the degree and timing of joint stiffness - 2 questions score 0-20). The WOMAC scores were normalized to a 0-100 point scale for data analysis, where 0 is no pain and higher scores indicate greater pain, stiffness or difficulty in performing daily tasks.
Time Frame: baseline, week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- AMZ001 BID: on the target knee
  AMZ001 gel twice daily.
- Placebo BID: on the target knee
  Placebo gel twice daily.
Arm/Group | AMZ001 BID | AMZ001 + Placebo QD | Placebo BID
Number analyzed (Participants) | 120 | 120 | 120
score on a scale
  Change from baseline WOMAC total score | -24.15 [-26.95 to -21.34] | -23.32 [-26.16 to -20.47] | -20.57 [-23.42 to -17.72]
  Change from baseline WOMAC function score | -23.43 [-26.29 to -20.58] | -22.30 [-25.19 to -19.40] | -19.94 [-22.84 to -17.04]
  Change from baseline WOMAC stiffness score | -23.17 [-26.42 to -19.93] | -23.35 [-26.66 to -20.05] | -20.65 [-23.96 to -17.34]

3. Secondary Outcome: WOMAC Pain Weight-bearing Score and Non-weight-bearing Score
Description: Change from baseline in Western Ontario McMasters Universities Osteoarthritis Index (WOMAC) pain weight-bearing score (questions 1,2, & 5; score 0-30) and non-weight-bearing score (questions 3&4; score 0-20) on target knee. The WOMAC scores were normalized to a 0-100 point scale for data analysis, where 0 is no pain and higher scores indicate greater pain, stiffness or difficulty in performing daily tasks.
Time Frame: baseline, week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | AMZ001 BID | AMZ001 + Placebo QD | Placebo BID
Number analyzed (Participants) | 120 | 120 | 120
score on a scale
  Change from baseline WOMAC pain weight bearing | -27.03 [-30.36 to -23.70] | -27.68 [-31.07 to -24.30] | -22.65 [-26.04 to -19.25]
  Change from baseline WOMAC pain non-weight bearing | -25.65 [-28.87 to -22.44] | -26.89 [-30.17 to -23.61] | -22.93 [-26.22 to -19.65]

4. Secondary Outcome: ICOAP Scores
Description: Change from baseline in Intermittent and Constant Osteoarthritis Pain (ICOAP) scores (score 0 [no pain]- 4 [extreme pain]). ICOAP scores were normalized to a 0-100 point scale, where 0 is no pain and higher scores indicate greater pain.
Time Frame: baseline, week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | AMZ001 BID | AMZ001 + Placebo QD | Placebo BID
Number analyzed (Participants) | 120 | 120 | 120
score on a scale
  ICOAP total score | -20.62 [-23.40 to -17.84] | -18.87 [-21.72 to -16.02] | -17.98 [-20.83 to -15.13]
  ICOAP constant pain score | -20.82 [-23.91 to -17.73] | -19.01 [-22.18 to -15.83] | -18.37 [-21.54 to -15.19]
  ICOAP intermittent pain score | -20.18 [-23.19 to -17.17] | -19.00 [-22.09 to -15.92] | -17.99 [-21.08 to -14.90]

5. Secondary Outcome: Physical Function
Description: Change in baseline in physical function assessed by the chair-stand test. The test measures the maximum number of chair stand repetitions possible in a 30-second period with out using the arms. Where 0 is no repetition completed and higher numbers corresponds to greater repetitions and physical function.
Time Frame: baseline, week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: repetitions
Arm/Group | AMZ001 BID | AMZ001 + Placebo QD | Placebo BID
Number analyzed (Participants) | 120 | 120 | 120
repetitions | 2.41 [1.98 to 2.83] | 2.30 [1.87 to 2.72] | 2.37 [1.94 to 2.80]

6. Secondary Outcome: Proportion of Responders as Per OMERACT-OARSI Criteria
Description: Outcome Measures in Rheumatology- Osteoarthritis Research Society International (OMERACT-OARSI) response involves changes that are deemed to be clinically relevant in three domains: pain, function, and PGA (Patient Global Assessment). For each of these domains, ranges are defined for absolute and percent changes from baseline that correspond to "high improvement" and "moderate improvement". OMERACT-OARSI response is defined as either high improvement in at least 1 of WOMAC pain and function scores OR moderate improvement in at least 2 of WOMAC pain scores, WOMAC function score or Patient Global Assessment (PGA)
Time Frame: week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of responders
Arm/Group | AMZ001 BID | AMZ001 + Placebo QD | Placebo BID
Number analyzed (Participants) | 115 | 109 | 109
Proportion of responders | 0.765 [0.679 to 0.834] | 0.826 [.0743 to 0.886] | 0.725 [0.634 to 0.800]

7. Secondary Outcome: Total Dose of Rescue Medication
Description: Total dose of rescue medication calculated as the average gram use/day, based on pill counts.
Time Frame: weeks 1 through 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: gram/day
Arm/Group | AMZ001 BID | AMZ001 + Placebo QD | Placebo BID
Number analyzed (Participants) | 120 | 120 | 120
gram/day | 0.27 [0.19 to 0.36] | 0.31 [0.22 to 0.40] | 0.30 [0.21 to 0.39]

8. Secondary Outcome: Time Between Baseline and First Use of Rescue Medication
Description: Time between baseline and first use of rescue medication.
Time Frame: weeks 1 through 4
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | AMZ001 BID | AMZ001 + Placebo QD | Placebo BID
Number analyzed (Participants) | 120 | 120 | 120
Days | 17 [7.0 to 24.0] | 9 [5.0 to 15.0] | 10 [4.0 to 17.0]

9. Secondary Outcome: WOMAC Pain Sub-score (Dose Comparison)
Description: Change from baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain sub-score (questions 1-5; score 0 [no pain]-50 [extreme pain]) on target knee. The WOMAC scores were normalized to a 0-100 point scale for data analysis, where 0 is no pain and higher scores indicate greater pain, stiffness or difficulty in performing daily tasks.
Time Frame: baseline, week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | AMZ001 BID | AMZ001 + Placebo QD
Number analyzed (Participants) | 120 | 120
score on a scale | -26.49 [-29.60 to -23.38] | -27.33 [-30.5 to -24.17]

10. Secondary Outcome: ICOAP Scores (Dose Comparison)
Description: as for outcome 4
Time Frame: baseline, week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | AMZ001 BID | AMZ001 + Placebo QD
Number analyzed (Participants) | 120 | 120
score on a scale | -20.62 [-23.40 to -17.84] | -18.87 [-21.72 to -16.02]

11. Secondary Outcome: WOMAC Pain Weight-bearing Score and Non-weight-bearing Score (Dose Comparison)
Description: Changes from baseline in Western Ontario and McMasters Universities Osteoarthritis Index (WOMAC) pain weight-bearing score (questions 1,2, & 5; score 0-30) and non-weight-bearing score (questions 3&4; score 0-20) on target knee. The WOMAC scores were normalized to a 0-100 point scale for data analysis, where 0 is no pain and higher scores indicate greater pain, stiffness or difficulty in performing daily tasks.
Time Frame: baseline, week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | AMZ001 BID | AMZ001 + Placebo QD
Number analyzed (Participants) | 120 | 120
score on a scale
  Weight-bearing | -27.03 [-30.36 to -23.70] | -27.68 [-31.07 to -24.30]
  Non-weight-bearing | -25.65 [-28.87 to -22.44] | -26.89 [-30.17 to -23.61]

12. Secondary Outcome: Physical Function (Dose Comparison)
Description: Change in baseline assessed by the chair-stand test. The test measures the maximum number of chair stand repetitions possible in a 30-second period with out using the arms. Where 0 is no repetition completed and higher numbers corresponds to greater repetitions and physical function.
Time Frame: baseline, week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: repetitions
Arm/Group | AMZ001 BID | AMZ001 + Placebo QD
Number analyzed (Participants) | 120 | 120
repetitions | 2.41 [1.98 to 2.83] | 2.3 [1.87 to 2.72]

13. Secondary Outcome: WOMAC Total Score and WOMAC Function and Stiffness (Dose Comparison)
Description: as for outcome 2
Time Frame: baseline, week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | AMZ001 BID | AMZ001 + Placebo QD
Number analyzed (Participants) | 120 | 120
score on a scale
  Function | -23.43 [-26.29 to -20.58] | -22.30 [-25.19 to -19.40]
  Stiffness | -23.17 [-26.42 to -19.93] | -23.35 [-26.66 to -20.05]

14. Secondary Outcome: Impact of Osteoarthritis on Daily Living (PGA Score)
Description: Change from baseline in Impact of OA daily living assessed using Patient Global Assessment (PGA) score. PGA is scored on a 11-point scale from 0 (none) to 10 (extreme), where higher scores represents a higher level of disease activity or worse health.
Time Frame: baseline, week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | AMZ001 BID | AMZ001 + Placebo QD | Placebo BID
Number analyzed (Participants) | 120 | 120 | 120
score on a scale | -2.29 [-2.63 to -1.94] | -2.31 [-2.66 to -1.96] | -1.68 [-2.03 to -1.32]

15. Secondary Outcome: Work Productivity
Description: Change from baseline in work productivity and activity assessed by the Work Productivity and Active Impairment (WPAI scores 0-100% in four different categories: absenteeism, presenteeism, work productivity loss, and activity impairment). Outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Time Frame: baseline, week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of impairment
Arm/Group | AMZ001 BID | AMZ001 + Placebo QD | Placebo BID
Number analyzed (Participants) | 45 | 41 | 39
percentage of impairment
  WPAI % Time missed | 0.39 [-2.73 to 3.51] | -3.10 [-6.43 to 0.23] | 1.58 [-2.01 to 5.16]
  WPAI % Impairment while working | -13.11 [-18.71 to -7.51] | -14.38 [-20.57 to -8.79] | -5.28 [-12.26 to 1.70]
  WPAI % Overall work impairment | -11.69 [-17.95 to -5.43] | -16.93 [-23.95 to -9.91] | -6.50 [-14.19 to 1.20]
  WPAI % Activity impairment | -17.75 [-21.45 to -14.06] | -20.41 [-24.15 to -16.68] | -13.03 [-16.79 to -9.27]

16. Secondary Outcome: Change in Quality of Life: EQ5D VAS Score
Description: The EuroQol-5 Domain (EQ-5D) is a standardized generic measure of health-related quality of life. The visual analog scale (VAS) is scored on a 0-100 scale, where 0 is "the worst health you can imagine" and 100, "the best health you can imagine".
Time Frame: baseline, week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | AMZ001 BID | AMZ001 + Placebo QD | Placebo BID
Number analyzed (Participants) | 120 | 120 | 120
score on a scale | 13.04 [10.13 to 15.94] | 11.76 [8.82 to 14.71] | 8.34 [5.39 to 11.28]

17. Other Pre Specified Outcome: Safety Endpoint (Adverse Events)
Description: Nature, incidence and severity of AEs.
Time Frame: weeks 1 through 4
Population: The SAF (Safety Analysis Set; N=121) was used for safety evaluation of adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | AMZ001 BID | AMZ001 + Placebo QD | Placebo BID | Voltaren 1% QID
Number analyzed (Participants) | 121 | 121 | 121 | 81
Participants
  All TEAEs | 51 | 53 | 75 | 26
  Deaths | 0 | 0 | 0 | 0
  SAEs | 0 | 0 | 0 | 0
  AEs leading to treatment discontinuation | 3 | 8 | 7 | 5
  ADR | 29 | 29 | 51 | 9
  Severity Mild | 39 | 45 | 66 | 20
  Severity Moderate | 17 | 11 | 14 | 9
  Severity Severe | 0 | 0 | 1 | 1

18. Other Pre Specified Outcome: Skin Tolerability Assessment (Skin Reactions)
Description: Skin tolerability assessment, incidence of erythema at the application site. Grading scheme from 0-4 (0, normal skin, no erythema; 4, blister formation and/or necrosis).
Time Frame: week 4
Population: Nature, incidence and severity of AEs. The SAF (Safety Analysis Set; N=121) was used for safety evaluation of adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | AMZ001 BID | AMZ001 + Placebo QD | Placebo BID | Voltaren 1% QID
Number analyzed (Participants) | 121 | 121 | 121 | 81
Participants
  Normal skin; no erythema | 100 | 89 | 79 | 68
  Questionable erythema not covering entire app site | 14 | 18 | 20 | 3
  Definite erythema not covering entire app site | 2 | 2 | 10 | 0
  Definite erythema and swelling or induration | 0 | 0 | 0 | 0
  Blister formation and/or necrosis | 0 | 0 | 0 | 1

19. Post Hoc Outcome: WOMAC Pain Sub-score (Subgroup With WOMAC Normalized Pain Sub-score ≥40 at Baseline)
Description: Change from baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain sub-score (questions 1-5; score 0 [no pain]-50 [extreme pain]) on target knee. The WOMAC scores were normalized to a 0-100 point scale for data analysis. The WOMAC scores were normalized to a 0-100 point scale for data analysis, where 0 is no pain and higher scores indicate greater pain, stiffness or difficulty in performing daily tasks.
Time Frame: baseline, week 4
Population: Post-hoc statistical analyses were performed for the comparison of each of the AMZ001 regimens vs placebo and between the two AMZ001 regimens. Sub-group of subjects meeting the WOMAC pain sub-score inclusion criterion at both screening and baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | AMZ001 BID | AMZ001 + Placebo QD | Placebo BID
Number analyzed (Participants) | 109 | 107 | 106
score on a scale | -28.54 [-31.87 to -25.20] | -29.02 [-32.45 to -25.60] | -23.18 [-26.64 to -19.72]

20. Post Hoc Outcome: WOMAC Total Score and WOMAC Function and Stiffness (Subgroup With WOMAC Normalized Pain Sub-score ≥40 at Baseline)
Description: Change from baseline in Western Ontario McMasters Universities Osteoarthritis Index (WOMAC) total score and WOMAC function (degree of difficulty experienced in performing daily activities - 17 questions score 0-170) and stiffness (the degree and timing of joint stiffness - 2 questions score 0-20) . The WOMAC scores were normalized to a 0-100 point scale for data analysis, where 0 is no pain and higher scores indicate greater pain, stiffness or difficulty in performing daily tasks.
Time Frame: baseline, week 4
Population: as for outcome 19
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | AMZ001 BID | AMZ001 + Placebo QD | Placebo BID
Number analyzed (Participants) | 109 | 107 | 106
score on a scale
  Change from baseline WOMAC total score | -25.54 [-28.54 to -22.54] | -24.03 [-27.11 to -20.95] | -20.61 [-23.71 to -17.51]
  Change from baseline WOMAC function score | -24.69 [-27.75 to -21.64] | -22.84 [-25.97 to -19.70] | -19.84 [-23.00 to -16.68]
  Change from baseline WOMAC stiffness score | -24.08 [-27.52 to -20.64] | -23.57 [-27.11 to -20.03] | -20.33 [-23.89 to -16.76]

ADVERSE EVENTS:
Time Frame: 4 Weeks
Arm/Group | AMZ001 BID | AMZ001 + Placebo QD | Placebo BID | Voltaren 1% QID
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/121 | 0/121 | 0/121
Serious Adverse Events (participants affected / at risk) | 0/121 | 0/121 | 0/121 | 0/121
Other Adverse Events (participants affected / at risk) | 29/121 | 30/121 | 52/121 | 11/81
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMZ001 BID (N=121) | AMZ001 + Placebo QD (N=121) | Placebo BID (N=121) | Voltaren 1% QID (N=81)
Headache (Nervous system disorders) | 2 (3) | 1 (2) | 8 (9) | 0 (0)
Application Site erythema (General disorders) | 11 (12) | 15 (16) | 40 (41) | 4 (4)
Application site dryness (General disorders) | 18 (18) | 13 (13) | 16 (16) | 5 (5)
Application site pruritus (General disorders) | 5 (5) | 8 (8) | 6 (6) | 2 (3)
Nasopharyngitis (Infections and infestations) | 6 (7) | 3 (3) | 6 (6) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/44/NCT03691844/SAP_000.pdf
  • Study Protocol (2018-11-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT03691844/Prot_001.pdf